CLINICAL TRIAL: NCT05348486
Title: FMISO-based Adaptive Radiotherapy for Head and Neck Cancer - a Prospective Multicenter Study
Brief Title: FMISO-based Adaptive Radiotherapy for Head and Neck Cancer
Acronym: FARHEAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Collaborators: Masaryk Memorial Cancer Institute (Other); University Hospital Ostrava (Other)
Responsible Party: Principal Investigator, Martin Dolezel, Profesor Martin Dolezel, M.D., Ph.D., University Hospital Olomouc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-03-00435
Record Dates: First submitted 2022-04-20; First posted 2022-04-27 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer; Hypoxia; FMISO; Dose Escalation
Keywords: Head and Neck Cancer; Hypoxia; Radiotherapy; Dose escalation
MeSH Terms: conditions — Head and Neck Neoplasms; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation (Experimental): Dose escalated radiotherapy protocol: 75,9 - 79,2 Gy in 33 fractions GTV hypoxic or any hypoxic LN > 2cm - PTV (0mm): dose 75,9 - 79,2 Gy/33 (Contours must be subtracted and reduce by 3mm in case of close relation to the skin, bones or large blood vessels) GTV primary - CTV - PTV (5+5mm): for dose 70 Gy/33 LN low risk (for elective irradiation) - CTV - PTV (3mm-5mm): for dose 54 Gy/33
  Interventions: Radiation: Dose escalation
- Standard fractionation (No Intervention): Standard fractionation regimen: 70 Gy/54 Gy in 33 fractions GTV primary - CTV - PTV (5+5mm): for dose 70 Gy/33 GTV LN bulky (> 3cm) - PTV (5mm): for dose 70 Gy/33 LN low risk (for elective irradiation) - CTV - PTV (3mm-5mm): for dose 54 Gy/33

INTERVENTIONS:
Radiation: Dose escalation — Dose escalation 75,9 - 79,2 Gy in 33 fractions for GTV hypoxic or any hypoxic LN > 2cm
  Arms: Dose escalation

SUMMARY:
Hypoxia occurs in about 80% of head and neck tumors. Based on experimental and clinical data, hypoxia is a useful parameter for pretherapeutic stratification. These radioresistant regions can be detected with FMISO PET/CT. Moreover, hypoxic subvolumes of tumors can be evolving as target volumes for radiotherapy ("dose painting") in hypoxia imaging-based dose escalation.

DETAILED DESCRIPTION:
The radiotherapy protocol will include two dose-escalation regimens. The dose in hypoxic tumor volume will be escalated either by conventional RT or stereotactic radiotherapy technique. Concurrent chemotherapy cisplatin will be administered weekly 35-40 mg/m2 or every three weeks 80-100 mg/m2. The parameter of cumulative cisplatin dose of 200 mg/m2 during the whole course of radiotherapy will be also taken into account. Patients will be examined and monitored at least every two weeks.

Target volumes and dose and fractionation:

Definition of gross tumor volumes (GTV), clinical target volumes (CTV) and planning target volumes (PTV) will follow recommendations of DAHANCA, EORTC and RTOG guidelines.

The conventional radiotherapy protocol:

Standard fractionation regimen: 70 Gy/54 Gy in 33 fractions GTV primary - CTV - PTV (5+5mm): for dose 70 Gy in 33 fractions GTV LN bulky (> 3cm) - PTV (5mm): for dose 70 Gy in 33 fractions LN low risk (for elective irradiation) - CTV - PTV (3mm-5mm): for dose 54 Gy in 33 fractions

Dose escalated radiotherapy protocol:

Dose escalated radiotherapy protocol: 75,9 - 79,2 Gy in 33 fractions GTV hypoxic or any hypoxic LN > 2cm - PTV (0mm): dose 75,9 - 79,2 Gy in 33 fractions (Contours must be subtracted and reduce by 3mm in case of close relation to the skin, bones or large blood vessels) GTV primary - CTV - PTV (5+5mm): for dose 70 Gy in 33 fractions LN low risk (for elective irradiation) - CTV - PTV (3mm-5mm): for dose 54 Gy in 33 fractions

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven new diagnosis of oropharyngeal p16 negative, or laryngeal, hypopharyngeal, oral cavity (independent of p16) squamous cell carcinoma of clinical stage III, IV confined to head and neck area
* Evaluable tumor burden assessed by computed tomography scan or magnetic resonance imaging, based on RECIST (Response Evaluation Criteria in Solid Tumours) version 1.1
* Eligibiity for definitive chemoradiation or hyperfractionated accelerated radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate kidney and liver function

Exclusion Criteria:

* Prior surgical treatment - any surgery of primary tumor or involved nodes or prior surgical debulking apart from surgery with diagnostic intention (e.g. open biopsy if necessary)
* Prior systemic therapy, targeted therapy, radiotherapy treatment for head and neck cancer
* Cancer outside of the oropharynx, larynx, and hypopharynx or oral cavity, such as nasopharyngeal, sinus, other para-nasal, or unknown primary head and neck cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis or any distant metastasis
* Known active Hepatitis B or C
* History of Human Immunodeficiency Virus (HIV)
* History of a diagnosed and/or treated hematologic or primary solid tumor malignancy, unless in remission for at least 5 years prior to randomization
* Previous allogeneic tissue/solid organ transplant
* Active infection requiring systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 2-year
  response rate
Locoregional progresion free survival | 2-year
  locoregional progresion free survival
Rate of acute (<3 months) radiation-induced events according to CTCAE 5.0 | 3 months
  acute radiation-induced events
Rate of late radiation-induced events according to CTCAE 5.0 | 2-year
  late radiation-induced events

SECONDARY OUTCOMES:
Overall survival | 4 years
  overall survival
Distant metastasis free survival | 4 years
  distant metastasis free survival
Change in QoL according to the standardised EQ-5D questionnaire | 2 years
  QoL according to the standardised EQ-5D questionnaire
Rate of new hypoxic areas after two weeks of radiotherapy | 2 week after start of radiotherapy
  rate of new hypoxic areas after two weeks of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dolezel, Prof., Principal Investigator — Palacký University and University Hospital Olomouc; Marek Slavik, Ph.D., Study Chair — The Masaryk Memorial Cancer Institute (MMCI); Jakub Cvek, Prof., Study Chair — Faculty Hospital Ostrava
Locations (3):
- Czechia (3):
  - The Masaryk Memorial Cancer Institute, Brno
  - Radiation oncology department in Palacký University and University Hospital Olomouc, Olomouc
  - Faculty Hospital Ostrava, Ostrava

IPD SHARING:
Plan to Share IPD: Undecided